CLINICAL TRIAL: NCT05408000
Title: Comparision of Motor Seizure Duration of Ketofol and Propofol for Electroconvulsive Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Dilip Baral, consultant Anesthesiologist, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1288
Record Dates: First submitted 2022-05-26; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Electroconvulsive Therapy
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketofol (Active Comparator): patient given titrated dose of ketofol
  Interventions: Drug: ketofol vs propofol
- propofol (Active Comparator): patient given titrated dose of propofol
  Interventions: Drug: ketofol vs propofol

INTERVENTIONS:
Drug: ketofol vs propofol — Patients planned for electroconvulsive therapy meeting the inclusion criteria and not having exclusion criteria will be randomized into two groups. Group K will receive titrated dose of Ketofol and Group P will receive titrated dose of Propofol for induction of anaesthesia
  Other Names: ketofol and propofol

SUMMARY:
Propofol is routinely used in our hospital for ECT. It causes hypotension and has anticonvulsant actions. Use of ketofol ( 1:1 combination of ketamine and propofol) during ECT can have longer seizure duration and better hemodynamics than propofol alone which ultimately leads to better therapeutic efficacy. Motor seizure duration of minimum 20-25 seconds is usually recommended for therapeutic efficacy of ECT.Patients planned for electroconvulsive therapy meeting the inclusion criteria and not having exclusion criteria will be randomized into two groups. Group K will receive titrated dose of Ketofol and Group P will receive titrated dose of Propofol for induction of anaesthesia

DETAILED DESCRIPTION:
Electroconvulsive therapy (ECT) is a common treatment method used in severe depression and other psychiatric diseases. Currently, most ECT procedures are carried out with muscle paralysis under general anesthesia. It is important to establish an accurate balance between adequate anesthesia depth and optimal seizure duration. The objective of anesthesia during ECT is to provide a rapid onset and balance of both unconsciousness and muscle relaxation for the duration of the electrical stimulus and subsequent seizure .Therefore, anesthetics that are used for general anesthesia during ECT should have rapid onset, rapid emergence, no interference with seizure activity and

longer seizure duration. A motor seizure lasting 20-25 seconds at minimum has been typically recommended for therapeutic efficacy of ECT . Common drugs used for ECT anesthesia are methohexital, thiopental, etomidate, propofol and ketamine. Methohexital exerts depressant action on seizure activity and is contraindicated in patients acute intermittent porphyria. Etomidate causes increased incidence of emesis. Similarly incidence of sinus bradycardia and premature ventricular contraction increased with the use of thiopental during ECT procedures .

For these reasons methohexital, thiopental and etomidate are not used in current anesthetic practice for electroconvulsive therapy Propofol as an anaesthetic in ECT has favorable characteristics such as rapid onset and emergence from anesthesia, minimal postoperative confusion and a lower incidence of hypertension or tachycardia during induction of anesthesia. However, it produces a dose- dependent decrease in seizure duration . Ketamine, is also used as an anesthetic agent in ECT because it has a favorable seizure inducing effect and increased seizure duration. But it is also not devoid of disadvantages. Its main disadvantages are that it produces hypertension, delayed recovery and precipitates psychomimetic emergence phenomena . So ketofol (1:1combination of ketamine and propofol) can be a good alternative to either propofol or ketamine used alone for anesthetic management for ECT. Ketamine mitigates propofol-induced hypotension, and propofol mitigates ketamine-induced vomiting and emergence agitation. Ketofol can also have better outcome on motor seizure duration than propofol alone. Therefore, the present study is designed to test the hypothesis that ketofol would be a good alternative anesthetic agent and better than propofol for ECT procedures.After obtaining approval from Institutional Review committee (IRC) of TUTH and Nepal health research council (NHRC) the process of enrolling the eligible patients into the study will be started. Patients will be assessed for eligibility. Patients meeting the inclusion criteria and not having the exclusion criteria will be enrolled in the study. Patients will be divided into two groups: Group P (propofol group,n=27) and Group K (ketofol group ,n=27) using computer generated random numbers. Blinding will be done by sealed envelope technique. Pre-anesthetic checkup will be conducted and a detailed history and complete physical examination will be done prior to procedure. Informed consent will be taken from the legal guardian of patient. Patient will be transferred to the pre anesthetic room. Baseline hemodynamic parameters (SBP, DBP, MAP, SPO2 and HR) will be taken and recorded. An 18 G IV cannula will be secured in appropriate hand of patient. Patient will be premedicated with glycopyrolate 0.2 mg 30 minutes prior to procedure. Patient will be transferred to operation theatre. III ECG leads, SPO2 probe and NIBP pressure cuff will be attached. Heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP) and oxygen saturation (SPO2) will

be continually monitored. Preoxygenation will be done via facemask at the rate of 5liter/min for 5 minutes. Anesthesia assistant will pick an envelope for each patient. Test solution will be prepared by anesthesia assistant as per the instructions in the envelope. Group K - In 10 ml syringe, 2ml of ketamine (50mg/ml solution) and 8ml of normal saline will be drawn to make the 10mg/ml solution of ketamine. Finally in another new 10 ml syringe 5ml of the freshly prepared solution of ketamine (10mg/ml) and 5ml of propofol (10mg/ml) will be mixed. The study drug thus prepared will contain 5mg /ml of propofol and 5mg / ml of ketamine. There will be two such 10ml syringe of ketofol. Group P - propofol (10mg/ml solution) will be drawn in labeled 10ml syringe. Two such 10ml syringes of propofol will be prepared. Patient in Group K will be administered an initial dose of 0.5mg/kg ketofol (0.25 mg/kg of propofol + 0.25 mg/kg of ketamine). Similarly, patient in Group P will be given an initial dose of 0.5mg/kg propofol. In both the group this initial dose will be given within 15 seconds. Five seconds after administration of drug, patient will be assessed for unresponsiveness to verbal commands (by calling patient's name) & loss of eyelash reflex. Then titrated dose of drug will be given at the rate of 1ml every 5 seconds until the patient no longer responds to verbal commands and there is loss of eyelash reflex. The required total dose of propofol or ketofol will be recorded. After loss of consciousness, hemodynamic parameters (SBP, DBP, MAP, HR & SPO2) will be taken and recorded. An isolated forearm technique will be performed by inflating the tourniquet in arm where the iv cannula is not placed. Then, succinylcholine, 1 mg/kg iv will be administered. Ventilation will be assisted with 100 % oxygen via face mask in all groups during the procedure. Bite block will be used prior to application of bifrontal electrodes.

Then a psychiatrist blinded to the study groups will administer electrical stimuli through bifrontal electrodes. The frequency will be set at 90Hz and current will be set at 800 milliampere.

The duration of the motor seizure will be defined as the time from the ECT stimulus to cessation of tonic-clonic motor activity in the 'isolated' arm. After the end of seizure, bite block will be removed and ventilation will be continued with 100% oxygen via face mask. The duration of motor seizures will be recorded. Hemodynamic parameters (SBP, DBP, MAP and HR) will be recorded 1mins and 5 mins after the end of seizure. Common complication encountered during

ECT are transient hypertension and tachycardia. Esmolol 5mg iv bolus will be given during such episodes. The time from the end of succinylcholine administration until spontaneous breathing, eye opening, and obeying commands will be recorded. Once the patient is awake, obeys commands and maintains oxygen saturation without supplemental oxygen, the patient will be transferred to postoperative room. Patient will be monitored with ECG, pulse oximeter and noninvasive blood pressure for one hour in postoperative room and then the patient will be transferred.

ELIGIBILITY:
Inclusion Criteria:

* • All patients scheduled for electroconvulsive therapy irrespective of ECT sessions.

  * Patients between 16 to 65 years of age
  * Patients with ASA -PS of I and II

Exclus• Pregnant patients

* Patients with a history of Epilepsy
* Patients taking any anticonvulsant medication
* Patients with a history of substance abuse or dependence
* Patients with a history of any adverse effect to any drugs used during the procedure

ion Criteria:

-

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Motor seizure duration | 20 to 25 seconds
  • To compare the duration of motor seizures between Ketofol and Propofol groups.

SECONDARY OUTCOMES:
• To compare the emergence time between the groups | 3 to 7 minutes
  eye opening, spontaneous breathing, obeys commands

CONTACTS AND LOCATIONS:
Overall Officials: Dilip Baral, Md, Principal Investigator — tuth; renu gurung, MD, Study Chair — tuth; hem raj paneru, MD, Study Chair — tuth; pankal joshi, MD, Study Chair — tuth
Locations (1):
- Dr Dilip Baral, Kathmandu, Bagmati Province, Nepal